CLINICAL TRIAL: NCT00540618
Title: A Phase II Randomized, Placebo-Controlled, Double-Blind Study of MEDI-507, A Humanized Monoclonal Antibody That Binds to the CD2 Receptor, Administered by Subcutaneous Injection to Adults With Plaque Psoriasis.
Brief Title: A Phase II Study of MEDI-507, Administered by Injection to Adults With Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP082
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — siplizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): MEDI-507
  Interventions: Drug: MEDI-507
- 2 (Placebo Comparator)
  Interventions: Other: Placebo
- 3 (Active Comparator): MEDI-507
  Interventions: Drug: MEDI-507
- 4 (Active Comparator): MEDI-507
  Interventions: Drug: MEDI-507

INTERVENTIONS:
Drug: MEDI-507 — Compare in a placebo controlled manner, the disease activity of three dosing regimens of MEDI-507 (Monoclonal Antibody)
  Arms: 1
Other: Placebo
  Arms: 2
Drug: MEDI-507 — Monoclonal Antibody (5 mg for 12 weeks and 5 mg for 6 weeks)
  Arms: 3
Drug: MEDI-507 — Administered 7 mg for 4 weeks by injection (Monoclonal Antibody)
  Arms: 4

SUMMARY:
To compare disease activity, as measured by PASI score, of three MEDI-507 dosing (injection)regimens vs. placebo.

DETAILED DESCRIPTION:
The primary objective of this study is to compare disease activity, as measured by PASI score, of three MEDI-507 dosing regimens (5 mg for 12 weeks, 5 mg for 6 weeks, 7 mg for 4 weeks) versus placebo administered weekly by SC injection.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis involving at least 10% of body surface area
* Age 18 through 65 years at the time of the first dose of study drug
* Both males and females are eligible. However, sexually active females, unless surgically sterile or at least 1 year post-menopausal, must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 30 days prior to the first dose of study drug and must agree to continue
* Currently receiving no therapy for psoriasis except emollients (certain other over-the-counter products may be allowed with prior approval of the sponsor)
* Written informed consent obtained from the patient
* Ability to complete follow-up period of 167 days as required by the protocol

Exclusion Criteria:

* Pustular, guttate, or erythrodermic psoriasis as the predominant disease type
* PASI score <8
* At screening (must be within 21 days before study entry) any of the following: lymphocyte count under 1,200 cells/mm3, WBC under 4,000 cells/mm3, hematocrit below 32%, platelets below 110,000 cells/mm3, creatinine, AST, ALT over 1.5 times upper limit of normal
* At screening (must be within 21 days before study entry) any clinical evidence of HIV, hepatitis B, hepatitis C or active hepatitis A infection
* Pregnancy (must have a negative serum pregnancy test within 21 days prior to the first dose of study drug, and urine pregnancy test must be negative on Study Day 0 before study entry)
* History of cancer (except excision of basal cell carcinoma)
* Any documented immunodeficiency
* A history of prior administration of monoclonal antibodies or related proteins
* Receipt of systemic retinoids, corticosteroids, cyclosporin A, methotrexate, phototherapy or coal tar treatment in the past 4 weeks
* Use of topical therapy (except emollients) for psoriasis in the past 2 weeks (certain other over-the-counter products may be allowed with prior approval of the sponsor)
* Receipt of any investigational drug therapy within 6 weeks before the first dose of study drug in this protocol (use of licensed agents for indications not listed in the package insert is permitted)
* Current or planned participation in a research protocol in which an investigational agent or therapy may be administered
* Nursing mother
* Acute illness including infections 15. Clinical manifestations of significant end organ dysfunction or failure that may compromise the safety of the volunteer in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2001-09; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Biological activity will be assessed primarily by the Psoriasis Activity and Severity Index (PASI) | Days 14, 28, 42, 56, 70, 91, 107, and 167

SECONDARY OUTCOMES:
Observe adverse and serious adverse events | Day 107 and 167

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Dingivan, M.D., Study Director — MedImmune LLC
Locations (43):
- United States (36):
  - MDS Pharma Services (US) Inc., Phoenix, Arizona
  - Bressinck-Parker-Dinehart-Sangster Dermatology, PA, Little Rock, Arkansas
  - Associates in Research, Inc., Fresno, California
  - nTouch Research Corporation, San Diego, California
  - Solano Clinical Research, Vallejo, California
  - Dermatology Specialists, Inc., Vista, California
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - Cherry Creek Dermatology, Denver, Colorado
  - The Savin Center, PC, New Haven, Connecticut
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - ICSL-Clinical Studies, Sarasota, Florida
  - Comprehensive Research Institute, Tampa, Florida
  - Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - Research Solutions, LLC, Evansville, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - FutureCare Studies, Springfield, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Medicine & Dentistry of New Jersey Robert Wood Johnson Medical School and Clinical Research Center, New Brunswick, New Jersey
  - Probe Inc., Riverside Park, New Jersey
  - Associates in Dermatology Research, Rutherford, New Jersey
  - Sadick Research Group, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University Dermatology Consultants, Inc., Cincinnatti, Ohio
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Northeast Clinical Research Center, Allentown, Pennsylvania
  - Paddington Testing Company, Philadelphia, Pennsylvania
  - Radiant Research, Philadelphia, Pennsylvania
  - Clinicalm Partners-LLC, Johnston, Rhode Island
  - Harmony Clinical Research, Inc., Johnson City, Tennessee
  - Dermatology Consultants, PC, Nashville, Tennessee
  - Veteran's Administration Medical Center, Nashville, Tennessee
  - Breco Research, Ltd., Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
- Canada (7):
  - The Dermatology Centre, Calgary, Alberta
  - NewLab Clinical Research, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Probity Medical Research, Waterloo, Ontario
  - Probity Medical Research, Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - International Dermatology Research, Montreal, Quebec